CLINICAL TRIAL: NCT06158295
Title: Effects of Walking Apnea at Low Lung Volume on Hypoalgesia, Cardiovascular Function and Respiratory Function
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Fran de Asís Fernández, Fran DeAsís-Fernández, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSEULS-PI-018/2023
Record Dates: First submitted 2023-11-18; First posted 2023-12-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pain; Hypoxia; Hypercapnia; Apnea
MeSH Terms: conditions — Pain; Hypoxia; Hypercapnia; Apnea

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking apnea at Low Lung Volume (Experimental): Participants walk at 5,5 km/h on treadmill for 6 minutes. Participants in the experimental group will perform intermittent apneas at low lung volume with a density of 15 seconds, followed by a normal breath of 10 seconds (15 cycles of 15s apnea - 10s normal breathing, until completing the 6 minutes).
  Interventions: Other: Voluntary apnoea
- Walking at normal breathing (No Intervention): Participants walk at 5,5 km/h on treadmill for 6 minutes. Participants in the control group will remain breathing normally for these 6 minutes.

INTERVENTIONS:
Other: Voluntary apnoea — Walking apneas at low lung volume
  Arms: Walking apnea at Low Lung Volume

SUMMARY:
The aim of this randomized controlled study is to explore the hypoalgesic response of a 6 minutes of intermittent walking apneas training session at low lung volume in healthy subjects; also, as secondary objectives, to analyze the cardiovascular and respiratory response produced during the intervention.

ELIGIBILITY:
Inclusion Criteria:

- Asymptomatic subjects aged between 18 and 64 years.

Exclusion Criteria:

* Cardiovascular, respiratory, metabolic, neurological or osteomuscular signs or pathologies.
* History of epilepsy.
* Pregnant
* Pharmacological treatment.
* Participants who present any type of pain on the day of the measurements or who have frequently suffered pain during the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold (PPT) on thumb, anterior tibial and spinous process of C7 | before and after intervention (up 30 minutes)
  PPT is tested on the dorsal base of the distal phalanx of the thumb on the dominant side and on the muscle belly of the tibialis anterior on the dominant side. The region to be pressed is marked with a pen. The patient is instructed to report with the first appearance of the sensation of "discomfort". An ascending ramp of 0.5 kg/cm/s is applied, at the rhythm of a metronome. The measurement is started on the thumb, and alternated with tibia and C7 until 3 measurements of each region are obtained, enough time to give 30 seconds of rest between measurements in the same region. This protocol has demonstrated high inter-observer reliability measuring healthy subjects (ICC = 0.91).

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | before intervention (up 5 minutes)
  14-item questionnaire about their thoughts and feelings in the last month. The scale has a range of scores from 0 to 56. The lower the score, the more favorable for the patient's health.
Pittsburg Sleep Quality Index (PSQI) | before intervention (up 5 minutes)
  9-item questionnaire on sleep quality in the past month. The scale has a range of scores from 0 to 21. The lower the score, the more favorable for the patient's health.
Global Physical Activity Questionnaire (GPAQ) | before intervention (up 5 minutes)
  6-item questionnaire on the level of physical activity at work, for commuting and in leisure time. A higher score means higher weekly physical activity.
Heart rate | during intervention (up 6 minutes)
  Heart rate will be measured during the procedure by finger pulse oximetry.
Oxygen saturation | during intervention (up 6 minutes)
  Oxygen saturation will be measured during the procedure by finger pulse oximetry.
Blood pressure | before, during and after intervention (up 10 minutes)
  Systolic and diastolic blood pressure will be measured before, during and immediately after the procedure using a digital wrist sphygmomanometer.
Rate of perceived exertion (RPE) | immediately after intervention (up 10 seconds)
  RPE Borg CR-10 is used to measure how hard your body works during physical activity. It runs from 0 - 10, using numbers to rate how much effort an activity takes.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU LaSalle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No